CLINICAL TRIAL: NCT04324541
Title: Health & Aging Brain Study: Health Disparities TAU Project
Status: Completed | Type: Observational
Sponsor: Sid E. O'Bryant (Other)
Responsible Party: Sponsor-Investigator, Sid E. O'Bryant, Executive Director, Institute for Translational Research Professor, Department of Pharmacology & Neuroscience, University of North Texas Health Science Center
Organization: University of North Texas Health Science Center (Other)
Other Study IDs: 2019-192
Record Dates: First submitted 2020-03-24; First posted 2020-03-27 (Actual); Results first posted 2024-05-17 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Brain Aging in Mexican Americans

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes

GROUPS / COHORTS (1):
- Mexican American Adults: No intervention
  Interventions: Diagnostic Test: PET scan of the brain with Flortaucipir

INTERVENTIONS:
Diagnostic Test: PET scan of the brain with Flortaucipir — PET scan of the brain with non FDA approved Radio tracer.

SUMMARY:
By doing this study we are trying to learn more about brain aging in Mexican Americans.

Participants will be asked to complete a screening visit to determine if it is safe to undergo a PET scan.

If eligible, participants will undergo a medical procedure that takes a picture of their brain. This procedure is called a PET scan of the brain.

ELIGIBILITY:
Inclusion Criteria:

* Participation in the Health & Aging Brain Study: Health Disparities Amyloid Project

Exclusion Criteria:

* Not a participant in the Health & Aging Brain Study: Health Disparites Amyloid Project
* Medical condition that precludes safe use of PET tracer

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Mexican Americans that participated in the Health & Aging Brain Study Amyloid Project
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2019-09-23 (Actual); Primary Completion 2019-10-17 (Actual); Study Completion 2021-04-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of North Texas Health Science Center Institute for Translational Research, Fort Worth, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Tau Scan Completed: Particiapnts completed screening and had Tau PET scan completed
Period: Overall Study
Arm/Group | Tau Scan Completed
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Tau Scan Completed: Participants completed screening and Tau PET scan
Arm/Group | Tau Scan Completed
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Tau Accumulation Measured by PET Imaging
Description: Tau PET scan completed and radiologist reviewed imaging and provided a report on whether or not Tau protein was present in the brain.
Time Frame: 4 weeks
Population: No analysis completed. Only aim was to complete Tau PET scans
Measure: Count of Participants; unit: Participants
Groups:
- Tau PET Scan Completed: The only measurement is that 12 participants had Tau PET scans completed.
Arm/Group | Tau PET Scan Completed
Number analyzed (Participants) | 12
Participants | 12

ADVERSE EVENTS:
Time Frame: 3 weeks, 3 days
Description: no adverse events occurred
Arm/Group | Mexican American Adults
All-Cause Mortality (participants affected / at risk) | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2019-09-13): https://cdn.clinicaltrials.gov/large-docs/41/NCT04324541/Prot_000.pdf